CLINICAL TRIAL: NCT00724594
Title: Safety of N-acetylcysteine in Maternal Chorioamnionitis
Brief Title: Safety of N-acetylcysteine in Maternal Chorioamnionitis (NAC in Chorio)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Dorothea D. Jenkins, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01NS052448 (NIH); R01NS052448 (NIH)
Record Dates: First submitted 2008-07-28; First posted 2008-07-29 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2021-04-12 (Actual); Status verified 2021-03

CONDITIONS: Chorioamnionitis; Brain Injury
Keywords: chorioamnionitis; maternal chorioamnionitis; neonatal white matter injury; N-acetylcysteine; NAC; anti-oxidant treatment
MeSH Terms: conditions — Chorioamnionitis; Brain Injuries | interventions — Acetylcysteine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-acetylcysteine (Experimental): Mother/infant pairs were stratified by gestational age into premature (P) and term (T) cohorts.
  Interventions: Drug: N-acetylcysteine
- Control (Active Comparator): Mother/infant pairs were stratified by gestational age into premature (P) and term (T) cohorts.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: N-acetylcysteine — NAC (100 mg/kg/dose) was given intravenously to mothers within 4 hours of diagnosis of chorioamnionitis, and every 6 hours until delivery. NAC was given to preterm (12.5 mg/kg/dose) and term infants (25 mg/kg/dose) every 12 hours for 5 doses after birth.
  Other Names: Acetadote, NAC
  Arms: N-acetylcysteine
Drug: Control — Saline was given in the same volume, at the same timing as NAC infusions
  Other Names: Saline
  Arms: Control

SUMMARY:
The purpose of this trial was to find the best dose of N-acetylcysteine (NAC) to decrease brain injury in babies exposed to intrauterine infection without causing significant side effects.

DETAILED DESCRIPTION:
Chorioamnionitits is an infection in the fluid and membranes surrounding the baby in utero. Intrauterine infection is associated with significant white and grey matter brain injury in newborns and is particularly important in the pathogenesis of periventricular leukomalacia (PVL) and cerebral palsy (CP). CP has been shown to be 4-9 times higher in babies exposed to intrauterine infection than in normal infants. Antibiotics have not changed the risk for brain injury in the newborn.

NAC is a promising anti-oxidant therapy that has shown effective neuroprotection in an animal model of chorioamnionitis, and has a favorable safety profile with limited and manageable side effects.

In this trial, intravenous NAC was given to mothers antenatally and to their infants postnatally, who presented with the diagnosis of chorioamnionitis, to evaluate safety and pharmacokinetics (PK) in mothers and infants. Mothers at ≥24 weeks gestation and their infants were randomized to receive either saline NAC within 4 hours of a clinical diagnosis of chorioamnionitis. Infants were stratified into term (≥ 33wk) and preterm (24-32wk) cohorts, due to different expected rates of metabolism and clearance.

Information gained from this trial will be used to determine how rapidly NAC is metabolized by mother, fetus, infant, and the ability of NAC to cross placenta. This study will also elucidate the safety of NAC in the setting of chorioamnionitis for fetal neuroprotection.

ELIGIBILITY:
Inclusion Criteria:

Participants had all of the following to qualify:

* Chorioamnionitis, defined as either 1) clinical diagnosis of choriomanionitis 2) maternal fever greater than or equal to 100 degrees F in the presence of rupture of membranes or 2 of the following: uterine tenderness, maternal WBC > 15,000 cells/mm, fetal tachycardia > 160 bpm, malodorous amniotic fluid, or in preterm group only, rupture of membranes and active preterm labor.
* Gestational age ≥ 24 completed weeks, by first trimester ultrasound or date of last menstrual period.
* No greater than 4 hours from onset of fever or diagnosis.

Exclusion Criteria:

Participants had none of the following:

* Asthma, steroid-dependent
* Clinical sepsis, whether viral or bacterial in nature, defined as fever with signs of cardiovascular compromise in mother (blood pressure < 90/50, heart rate > 120 bpm, need for oxygen due to maternal saturations below 92%, pneumonia, pyelonephritis, or meningitis)
* Seizure disorder
* Fetal weight or biparietal diameter less than the 10th% for gestational age
* Suspected major genetic or congenital abnormality
* Fetal distress which demands immediate delivery (poor fetal biophysical profile, late decelerations, sinusoidal fetal heart rate pattern)
* Participation in another therapeutic clinical trial

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-08; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothea D. Jenkins, MD, Principal Investigator — Medical University of South Carolina; Eugene Chang, MD, Principal Investigator — Medical University of South Carolina (Obstetric Principal Investigator)
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Result] Wiest DB, Chang E, Fanning D, Garner S, Cox T, Jenkins DD. Antenatal pharmacokinetics and placental transfer of N-acetylcysteine in chorioamnionitis for fetal neuroprotection. J Pediatr. 2014 Oct;165(4):672-7.e2. doi: 10.1016/j.jpeds.2014.06.044. Epub 2014 Jul 23. PMID 25064164
- [Derived] Jenkins DD, Wiest DB, Mulvihill DM, Hlavacek AM, Majstoravich SJ, Brown TR, Taylor JJ, Buckley JR, Turner RP, Rollins LG, Bentzley JP, Hope KE, Barbour AB, Lowe DW, Martin RH, Chang EY. Fetal and Neonatal Effects of N-Acetylcysteine When Used for Neuroprotection in Maternal Chorioamnionitis. J Pediatr. 2016 Jan;168:67-76.e6. doi: 10.1016/j.jpeds.2015.09.076. Epub 2015 Nov 3. PMID 26545726

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due two enrolling two sets of twins (one set in the preterm/NAC group, and one set in the preterm/control group), our study included 24 infants and 22 mothers.
Groups:
- NAC Infant: Infants treated with N-acetylcysteine
- Control Infant: Infants treated with saline
- NAC Maternal: Mothers of infants treated with N-acetylcysteine
- Control Maternal: Mothers of infants treated with saline
Period: Overall Study
Arm/Group | NAC Infant | Control Infant | NAC Maternal | Control Maternal
Started | 12 | 12 | 11 | 11
Completed | 12 | 12 | 11 | 10
Not Completed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NAC Infant | Control Infant | NAC Maternal | Control Maternal | Total
Number analyzed (Participants) | 12 | 12 | 11 | 11 | 46
Age, Customized [Number; unit: participants]
  Preterm Infants | 7 | 7 | NA — Only applicable to infants | NA — Only applicable to infants | NA — Total not calculated because data are not available (NA) in one or more arms.
  Term Infants | 5 | 5 | NA — Only applicable to infants | NA — Only applicable to infants | NA — Total not calculated because data are not available (NA) in one or more arms.
  Mothers aged 18-45years | NA — Only applicable to mothers | NA — Only applicable to mothers | 11 | 11 | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11 | 11 | 33
  Male | 7 | 6 | 0 | 0 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 5 | 8 | 4 | 26
  White | 3 | 7 | 3 | 7 | 20
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 11 | 11 | 46

OUTCOME MEASURES:

1. Primary Outcome: NAC Terminal Elimination Half-life
Time Frame: prior to delivery in mothers, and in newborn after delivery during 2 days of NAC infusion
Measure: Mean (Standard Deviation); unit: hours
Groups:
- NAC Maternal: Mothers treated with N-acetylcysteine prior to delivery of infant
- NAC Preterm Infants: Preterm infants treated with N-acetylcysteine
- NAC Term Infants: Term infants treated with N-acetylcysteine
Arm/Group | NAC Maternal | NAC Preterm Infants | NAC Term Infants
Number analyzed (Participants) | 11 | 7 | 5
hours | 1.2 (0.2) | 7.5 (2.0) | 5.1 (1.3)

2. Primary Outcome: NAC Volume of Distribution
Time Frame: prior to delivery in mothers, and in newborn after delivery during 2 days of NAC infusion
Measure: Mean (Standard Deviation); unit: L/kg
Arm/Group | NAC Maternal | NAC Preterm Infants | NAC Term Infants
Number analyzed (Participants) | 11 | 7 | 5
L/kg | 0.41 (0.07) | 0.47 (0.04) | 0.38 (0.09)

3. Primary Outcome: NAC Total Body Clearance
Time Frame: prior to delivery in mothers, and in newborn after delivery during 2 days of NAC infusion
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | NAC Maternal | NAC Preterm Infants | NAC Term Infants
Number analyzed (Participants) | 11 | 7 | 5
mL/h/kg | 255 (61) | 45.0 (8.2) | 53.7 (11.3)

4. Primary Outcome: NAC Concentrations
Time Frame: Peak: 30 minutes after NAC infusion. Cord: at delivery
Measure: Mean (Standard Deviation); unit: micromol/L
Groups:
- NAC Maternal: Mothers treated with N-acetylcysteine prior to delivery
Arm/Group | NAC Maternal | NAC Preterm Infants | NAC Term Infants
Number analyzed (Participants) | 11 | 7 | 5
micromol/L
  Peak NAC concentration in plasma | 1222 (415) | 49.0 (14.9) | 92.3 (69.2)
  NAC cord concentration | NA (NA) — Not applicable to mothers | 370.7 (199.2) | 639.7 (409.4)

5. Primary Outcome: Placental Transfer Ratio
Description: Ratio of NAC concentration in cord to maternal venous blood
Time Frame: At time of delivery
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- NAC Maternal: Mothers treated with N-acetylcysteine prior to birth
Arm/Group | NAC Maternal
Number analyzed (Participants) | 12
ratio | 1.4 (0.8)

6. Primary Outcome: Maternal and Infant Mean Blood Pressure Change
Time Frame: Maternal mean BP changes were pre/post dosing prior to delivery. Infant measurements were pre/post their first dosing
Population: The infant and maternal populations analyzed for this portion are incomplete, as not all individuals had paired before/after blood pressure measurements at this time point.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- NAC Infants: Infants treated with N-acetylcysteine
- Control Infants: Infants treated with saline
- Control Maternal: Mothers treated with saline prior to delivery
Arm/Group | NAC Infants | Control Infants | NAC Maternal | Control Maternal
Number analyzed (Participants) | 10 | 7 | 11 | 10
mmHg | -1.2 (13) | 2.1 (11) | 1 (12) | 2 (10)

7. Primary Outcome: Cerebral Blood Flow
Description: Resistive index in middle cerebral artery (MCA)
Time Frame: after NAC infusion
Population: blood flow resistive indices after first dose of N-acetylcysteine or saline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Control Term Infants: Term Infants treated with saline
- Control Preterm Infants: Preterm Infants treated with saline
Arm/Group | NAC Term Infants | Control Term Infants | NAC Preterm Infants | Control Preterm Infants
Number analyzed (Participants) | 5 | 4 | 6 | 5
units on a scale | 0.93 [0.87 to 0.99] | 0.89 [0.81 to 0.97] | 0.92 [0.88 to 0.97] | 0.89 [0.82 to 0.95]
Statistical Analysis 1: Comparison: NAC Term Infants vs Control Term Infants; Term infant cohort : NAC vs control H0= there will be no difference in resistive index in Middle Cerebral Artery after N-acetylcysteine or saline in the term cohort; Test type: Other; p = 0.9, t-test, 2 sided — not significant
Statistical Analysis 2: Comparison: NAC Preterm Infants vs Control Preterm Infants; Preterm infant cohort: NAC vs control H0= there will be no difference in resisitive index in MCA after N-acetylcysteine or saline in preterm cohort; Test type: Other; p = 0.9, t-test, 2 sided

8. Primary Outcome: Prothrombin Time
Description: prothrombin clotting time
Time Frame: after N-acetylcystiene or saline infusion
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | NAC Infant | Control Infant | NAC Maternal | Control Maternal
Number analyzed (Participants) | 8 | 6 | 11 | 11
seconds | 19.5 (2.5) | 19.0 (4.0) | 14.2 (0.6) | 14.4 (1.2)
Statistical Analysis 1: Comparison: NAC Maternal vs Control Maternal; Maternal cohort: NAC versus control l H0= PT will not be different in mothers after NAC or saline; Test type: Other; p = 0.9, t-test, 2 sided — not significant
Statistical Analysis 2: Comparison: NAC Infant vs Control Infant; Infant cohort: NAC versus control H0= prothrombin time will not be different in the infants after NAC or saline; Test type: Other; p = 0.9, t-test, 2 sided

9. Secondary Outcome: Magnetic Resonance Spectroscopy of Infants
Description: ratio of myoInositol / NAA concentrations in basal ganglia
Time Frame: 36 - 40 weeks gestational age
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | NAC Infants | Control Infants
Number analyzed (Participants) | 7 | 9
ratio | 1.09 (0.31) | 1.34 (0.20)
Statistical Analysis 1: Comparison: NAC Infants vs Control Infants; correcting for gestational age at birth; Test type: Other; p = 0.072, t-test, 2 sided

10. Secondary Outcome: Cytokine Level IL-1Ra in Plasma
Description: anti-inflammatory cytokine Interleukin -1 Receptor alpha (IL-1Ra)
Time Frame: after N-acetylcysteine infusion
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | NAC Infants | Control Infants
Number analyzed (Participants) | 12 | 9
pg/ml | 745 [251 to 1302] | 8.3 [8.3 to 448]
Statistical Analysis 1: Comparison: NAC Infants vs Control Infants; Test type: Other; p = 0.014, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Mothers were monitored for Adverse Events for up to 2 days after treatment. Infants were assessed for Adverse Events until discharge, Serious Adverse Events up to 30 days post-treatment.
Arm/Group | NAC Infant | Control Infant | NAC Maternal | Control Maternal
Serious Adverse Events (participants affected / at risk) | 4/12 | 3/12 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 5/12 | 3/12 | 2/11 | 2/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAC Infant (N=12) | Control Infant (N=12) | NAC Maternal (N=11) | Control Maternal (N=11)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Resuscitation-chest compressions/CV meds
IVH 1-2 days of age (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
IVH 5-7 days of age (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
NEC within 30 days (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxic Ischemic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Culture Proven Sepsis (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | NAC Infant (N=12) | Control Infant (N=12) | NAC Maternal (N=11) | Control Maternal (N=11)
Rash/Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shortness of breath/wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Prolonged PT time (Blood and lymphatic system disorders) | 5/8 (5) | 3/6 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No